CLINICAL TRIAL: NCT02800395
Title: Influence of Oxidative Stress and Nutrition Biomarkers on the Cognitive Decline Evolution in Alzheimer Disease
Acronym: GERIOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014.860
Record Dates: First submitted 2016-05-30; First posted 2016-06-15 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; oxydative stress; nutrition; biomarkers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutritional evaluation (Other)
  Interventions: Procedure: Malnutrition screening and perioperative nutritional support

INTERVENTIONS:
Procedure: Malnutrition screening and perioperative nutritional support — * Multidisciplinary training sessions for malnutrition and malnutrition risk screening, postoperative nutritional procedures according to the ESPEN Guidelines
  * Preoperative Geriatric evaluation : eligibility criteria, nutritional status, previous history, comorbidities, clinical examination, activities of daily living (ADL) and Instrumental activities of daily living (IADL)
  * Implementation of an adapted nutritional support based on ESPEN Guidelines

SUMMARY:
According to several reports, the oxidative stress and the nutrition could have an impact in the Alzheimer disease.

The association of these two parameters measurements and the cognitive impairment decline could help in a predictive diagnosis of cognitive decline evolution in patients presenting cognitive disorders.

This is a monocentric prospective "routine care" clinical trial on patients showing cognitive troubles especially memory complaints.

The objective is to demonstrate a correlation between oxydative stress and nutrition biomarkers and the clinical evolution of patients complaining of cognitive impairments.

The neuropsychologic data collection (the mini mental Status Examination (MMSE), the clock test, the Grober-Buschke test (FCSR-IR), the executive function evaluated by the Trail making test, and the medical imaging (by magnetic resonance imaging (MRI) or tomography in case of MRI contraindication) will be realized during the study inclusion phase in the usual intake of patients. Whole blood samples for the oxydative and nutrition biomarkers measurements will be taken at the study inclusion day during the stay at the Day hospital dedicated to the routine intake of patients issued from the memory consultation.

In this study, the principal evaluation criteria will be the MMSE score evolution during the 60 months of the patients follow-up, measured during the routine visits scheduled approximately every 6 months, according to the french national authority for health recommendations. It will allow evaluating the correlation between the cognitive decline evolution measured by MMSE during the Alzheimer disease or related diseases method during the 2 years follow-up, and the oxydative stress blood markers.

ELIGIBILITY:
Inclusion Criteria:

* >55 years old patient
* Patient seen during a memory consultation in geriatric Unit, Lyon Sud University Hospital
* Patient or legal representative and/or person of confidence who didn't express his opposition to the clinical assay participation.
* Patient registered to the general social insurance
* Complementary health check scheduled at day hospital, conventional hospitalization or regular consultation.

Exclusion Criteria:

* Patient unable to express his participation refusal and under curatorship or unforced by the court of justice

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2014-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change (evolution) of patient's cognitive profile evaluation measured by MMSE score method during memory consultation follow-up, every 6 months until patient loss. | at baseline (day 0) and at 6, 12, 18, 24, 30, 36, 42, 48 months
  Patient cognitive profile evolution measured by successive MMSE score evaluations during follow-up memory consultation, every 6 months until patient loss.

SECONDARY OUTCOMES:
cognitive profile evaluation at inclusion phase | at baseline (day 0)
  Dubois's "5 words" test; free recall test; cued recall memory test; Trail Making Test Part A/Trail Making Test Part B (TMTA/TMTB)
Présence of cardiovascular risk factor | at baseline (day 0)
  arterial hypertension; Tobacco: estimated consumption in cigarettes pack per year; lipidemia: cholesterol, high-density lipoprotein cholesterol (HDLc), Triglycerides, low-density lipoprotein cholesterol (LDLc); diabetes: diabetes fasting blood glucose, HbA1c; prior cardiovascular histories: acute coronary syndrome, arteriopathy
treatment evaluation | at baseline (day 0) and at 6, 12, 18, 24, 30, 36, 42, 48 months
  drugs list, posology, indication Drug type (ACE inhibitors; NSAIDs; statins…) angiotensin-converting-enzyme inhibitor (ACE inhibitor) Nonsteroidal anti-inflammatory drugs (usually abbreviated to NSAIDs)
Functionality | at baseline (day 0) and at day hospital visit if need be (up to 48 months)
  Katz and Lawton scores ( ADL/ IADL)
Presence of anomalies on cerebral imaging data that evoke neuro-degenerative pathology, by MRI | At day hospital visit if need be (up to 48 months)
  Description: cortical atrophy; specific hippocampus cortex atrophy ( according to Sheltens classification); subcortical atrophy; vascular Leukoencephalopathy symptoms on T2-FLAIR sequence; micro-bleeds in T2 sequence; Iron deposition observed by MRI method (or CT scans if MRI is contraindicated)

CONTACTS AND LOCATIONS:
Overall Officials: Marc BONNEFOY, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Médecine Gériatrique. Groupement Hospitalier Sud. Hospices Civils de Lyon., Pierre-Bénite, France